CLINICAL TRIAL: NCT03160599
Title: Restricted Calorie Ketogenic Diet as a Treatment in Glioblastoma Multiforme: a Clinical Study
Brief Title: Restricted Calorie Ketogenic Diet as a Treatment in Malignant Tumors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCYY
Record Dates: First submitted 2017-05-02; First posted 2017-05-19 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Malignant Tumors
MeSH Terms: conditions — Neoplasms | interventions — Diet, Ketogenic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Restricted Calorie Ketogenic Diet (Experimental): Calorie restriction: The basis of dietary design is 70-85% of individual's total calories. The total calorie is based on patient's activity level and their basal metabolism values, which is obtained from indirect calorimetry or harris-benedict formula.
  Treatment will consist of ketogenic diet. KD will consist of 4:1-1:1[fat]:[protein+carbohydrate].Carbohydrate is limited to 10-30 g / day.The diet will be supplemented with vitamins, calcium, phosphorus, zinc and selenium supplements to meet the requirements of US Dietary Reference Intakes (DRI) standard.
  Interventions: Other: ketogenic diet

INTERVENTIONS:
Other: ketogenic diet — The treatment is mainly restricted calorie ketogenic diet. KD will consist of 4:1-1:1[fat]:[protein+carbohydrate].Carbohydrate is limited to 10-30 g / day.

SUMMARY:
Malignant tumor incidence showed an upgrade trend in recent years. Standard therapy for malignant tumor includes surgery followed by radiation and chemotherapy. Despite optimal treatment the prognosis remains poor. There is an urgent need for more effective therapies. The Warburg effect has been widely observed in human cancers. The main energy supply of tumor cells are aerobic glycolysis. Therefore, they are highly dependent on glucose metabolism. Recently, some scholars have suggested that 'Restricted calorie Ketogenic Diet (RKD)' might be able to inhibit glycolysis and thus anti-tumor by restricting carbohydrate intake. This will 'starve' cancer cells, which will lead to cell death. There are many animal and in vitro studies shown that RKD can reduce the tumor size and thus tumor cell growth of malignant tumors. However, a consistent positive result can not be found within a small sample of clinical trials. In this study, 40 patients with malignant tumors will be treated with or without RKD. The safety and efficacy of RKD and the patients' tolerance will be observed in order to understand whether this therapy can be a potential new treatment This clinical study is comparatively large internationally. It is the first domestically. This study is essential to extend the survival of patients with malignant tumors, and to study clinical nutrition support and its metabolic pathways for malignant tumors.

ELIGIBILITY:
Inclusion Criteria:

1. 40 patients with diagnosed/recurrent malignant tumors
2. Ability and willingness to sign informed consent form.

Exclusion Criteria:

1. Anticoagulation treatment with coumadin≥ 1 mg/day for ≤ 7 days prior to screening (low-dose [≤ 1 mg/day] coumadin, heparin, and low-molecular-weight heparin are permitted)
2. Any systemic illness or unstable medical condition that might pose additional risk, including: cardiac, unstable metabolic or endocrine disturbances, renal or liver disease, past history of renal calculi, hyperuricemia, hypercalcemia, mitochondrial disease, known disorder of fatty acid metabolism, porphyria, carnitine deficiency and pancreatitis
3. History of malignant tumors other than malignant glioma, such as surgical resection of non-melanoma skin cancer or cervical carcinoma in situ.
4. History of uncontrollable hyperlipidemia.
5. Active drug or alcohol dependence or any other factors that, in the opinion of the site investigators, would interfere with adherence to study requirements
6. History of having human immunodeficiency virus, or hepatitis C
7. Failure to recover from <CTCAE grade 2 toxicities related to prior therapy
8. Pregnancy or breastfeeding.
9. Use of any investigational drug within 1 months of enrollment
10. Inability or unwillingness of subject to give written informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events of patients on high-fat diet | 2 year
  The main focus of this period is to recruit patients and collect clinical data for patients with glioblastoma multiforme on restricted calorie ketogenic diet. The safety and tolerability of the treatment will be evaluated.This can be measured by reports of adverse incidences.

CONTACTS AND LOCATIONS:
Locations (1):
- the Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol